CLINICAL TRIAL: NCT01839760
Title: Prospective Study to Evaluate Viral Shedding Patterns and Clinical Outcomes of Hospitalized Adult Influenza Patients
Brief Title: Evaluation of Viral Shedding Patterns and Clinical Outcomes of Influenza Patients
Status: Completed | Type: Observational
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Other Study IDs: FLU-EPI-001
Record Dates: First submitted 2013-04-08; First posted 2013-04-25 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Viral shedding; Epidemiology
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inpatient cohort: Patients admitted to general wards
- ICU cohort: Patients admitted to ICU

SUMMARY:
The objective of the study is virological assessment (e.g., proportion of prolonged viral shedding, median days to viral clearance, and viral load) in laboratory-confirmed adult influenza patients admitted to the general ward and/or to the ICU and to assess the correlation with the clinical manifestations and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Hospitalized or admitted to ICU for influenza
* Age ≥18 years
* Laboratory confirmation of influenza A or B

Exclusion Criteria:

* Informed consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with laboratory-confirmed influenza A or B
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Viral load/Viral shedding | Day 7
  Outcome is the decay rate in viral load during hospital stay measured by quantitative polymerase chain reaction (QPCR)
Viral load/Viral shedding | Day 9
  Outcome is the decay rate in viral load during hospital stay measured by quantitative polymerase chain reaction (QPCR)
Viral load/Viral shedding | Day 11
  Outcome is the decay rate in viral load during hospital stay measured by quantitative polymerase chain reaction (QPCR)
Viral load/Viral shedding | Day 13
  Outcome is the decay rate in viral load during hospital stay measured by quantitative polymerase chain reaction (QPCR)
Viral load/Viral shedding | Day 15
  Outcome is the decay rate in viral load during hospital stay measured by quantitative polymerase chain reaction (QPCR)

CONTACTS AND LOCATIONS:
Locations (5):
- Northwestern University, Chicago, Illinois, United States
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario